CLINICAL TRIAL: NCT05669352
Title: A Phase 1/2 Study of Oral IRAK-4 Inhibitor CA-4948 in Combination With Pembrolizumab and Stereotactic Radiosurgery in Patients With Melanoma Brain Metastases
Brief Title: A Study of Oral IRAK-4 Inhibitor CA-4948 in Combination With Pembrolizumab and Stereotactic Radiosurgery in Patients With Melanoma Brain Metastases
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: uncertain study staffing
Sponsor: University of Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UF-CUT-002
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Melanoma Metastatic in the Brain
Keywords: melanoma; stereotactic radiosurgery; brain metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — CA-4948; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CA-4948 and Pembrolizumab (Experimental)
  Interventions: Drug: CA-4948; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CA-4948 — Subjects on both the phase I and phase II portions will take 200 mg CA-4948 orally two times daily.
Drug: Pembrolizumab — Subjects on both the phase I and phase II portions will receive 400 mg pembrolizumab intravenously once every six weeks.

SUMMARY:
This phase I/II trial will investigate the use of the novel oral IRAK-4 inhibitor CA-4948 in combination with pembrolizumab therapy following stereotactic radiosurgery (SRS) in patients with melanoma brain metastases (MBM). The investigators hypothesize that the addition of CA-4948 will reduce the rate of distant intracranial failure and reduce the need for subsequent radiation therapy. The investigators also propose that it will have a significant reduction in radiation necrosis and improve patient-reported symptoms and quality of life. This trial represents the first time an oral IRAK-4 inhibitor has been used in combination with aPD1 therapy in MBM and will yield valuable insight into its synergistic potential both in MBM and additional sites of metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiographic or histologically confirmed melanoma brain metastases (MBM) and be planning to undergo or have undergone SRS for treatment
* Patients must have measurable disease
* Patients may be treatment-naïve or currently on therapy for systemic disease control at time of MBM development. If MBM diagnosis coincides with initial diagnosis, patients may be treatment-naïve with systemic disease.

In patients naïve to treatment, the choice of initial therapy will be left up to the treating physician. If in their clinical judgement, single agent aPD1 plus SRS is deemed the appropriate therapy then these patients may proceed to enrollment and inclusion of CA-4948 with their regimen. If in the treating physician's judgement, patient would benefit from use of combination immunotherapy with CTLA-4/aPD1 therapy, then patient must complete induction with CTLA-4/aPD1 therapy and proceed to maintenance aPD1 therapy prior to enrollment. The timing of SRS in these patients should coincide with the conclusion of induction dual agent therapy (either during or following last cycle of CTLA-4/aPD1 therapy) to then allow for a 3-week washout from last dose of CTLA-4 inhibitor exposure received prior to starting on study drug with CA-4948 and pembrolizumab.

* Completion of induction is defined as either completing the planned 4 doses of CTLA-4/aPD1 therapy or if the CTLA-4 inhibitor is discontinued after any of the initial 3 doses of therapy due to toxicity. In the event for stopping due to toxicity, then patients may still be eligible for study inclusion as long as this toxicity would not prevent them from continuing on aPD1 therapy as planned systemic treatment and no other rules for exclusion have been met below. In these patients, the timing of SRS should be consistent as above and the washout period from time of last CTLA-4 inhibitor must be at least 3 weeks prior to initiating on study drug. If a longer period of washout is required due to toxicity and safe resumption of immunotherapy, patients may still be enrolled as long as they meet the timing requirements from time of SRS to initiation of therapy as outlined below.

  * In patient who develop MBM while previously having received treatment for metastatic melanoma at other systemic locations, previous treatment with dual checkpoint inhibitor therapy (CTLA-4/aPD1 or LAG-3/aPD-1) or single agent immunotherapy therapy will be allowed, as long as at the time of SRS to these MBM lesions the patient is planned to receive aPD1 therapy as long as the above criteria are met and the patients systemic disease is displaying at least SD on last surveillance imaging performed.
  * SD is determined by clinician judgement at time of study enrollment. In patients on systemic single agent aPD1 there is no washout necessary in this case and patients can start pembrolizumab and study drug at next scheduled cycle of treatment following completion of SRS as long as all other rules have been met for enrollment.
  * Previous oral BRAFi/MEKi treatment will also be allowed, as long as at the time of MBM treatment with SRS the patient is planned to initiate aPD1 therapy and not continue on BRAFi/MEKi. A washout period of 14 days from last dose of BRAFi/MEKi to initiation of study drug is required.
  * Treatment of symptomatic MBM with corticosteroids is allowed while receiving CA- 4948, but in order to start aPD1 therapy, patient must be on ≤ 10mg of oral prednisone daily or equivalent.

    * Patients must be tolerant of receiving MRI and cannot have intolerance to gadolinium contrast.
    * Age ≥18 years at time of informed consent.
    * ECOG performance status ≤1
    * Patients must have adequate organ and marrow function as defined below:
* absolute neutrophil count ≥ 1,500/mcL
* platelets ≥ 100,000/mcL
* hemoglobin ≥ 9.0 g/dL or ≥5.6 mmol/L
* coagulation PT/INR and aPTT ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic ranged of intended use for anticoagulants
* total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) OR direct bilirubin no lower than the ULN if total bilirubin > 1.5 × ULN
* AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN (with confirmed liver metastases: AST and ALT ≤ 5 x ULN)
* creatinine clearance (CrCl)≤ 1.5 × ULN measured or calculated OR glomerular filtration rate (GFR)≥ 30 mL/min based on modified Cockcroft and Gault formula for participants with creatinine levels > 1.5 × institutional upper limit of normal (ULN)

  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
  * Participants who are HBsAg positive are eligible if they have received hepatitis B antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization. Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
  * Subjects of childbearing potential must have a negative serum pregnancy test at screening and agree to use of highly effective methods of contraception throughout the study and for at least four months following the last dose of study treatment.
  * Subjects with partners of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation and 4 months after completion of CA-4948 administration. Subjects should also not donate sperm from first dose of therapy until 4 months after the last dose of treatment.
  * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
  * Participants must have recovered from all adverse events due to previous therapies to ≤Grade 1 or baseline with the exception of alopecia. Participants with ≤Grade 2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
  * Archival tumor tissue sample or newly obtained biopsy of a tumor lesion not previously irradiated has been provided.
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subject of child-bearing potential who has a positive urine pregnancy test within 72 hours prior to treatment
* Subject has received prior systemic anti-cancer therapy including investigational agents or devices within 4 weeks prior to screening
* If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
* Prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids over ≤ 10mg of oral prednisone daily or equivalent, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed. mRNA COVID-1 vaccines are allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab, CA-4948, or any of their excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of non-infectious pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy, is patient is receiving oral antibiotics for localized infection with planned end date they may enroll on study as soon as duration is complete.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the trial's requirements.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* Unable to discontinue medications contraindicated to CA-4948 or pembrolizumab.
* Patients with uncontrolled intercurrent illness.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reduction in need for repeated intercranial intervention 1 year after initial stereotactic radiosurgery (SRS) | 1 year
  Determine if the combination of CA-4948 and pembrolizumab reduces the need for repeated intercranial intervention 1 year after initial SRS, as measured by remaining free from need for repeated intracranial intervention 1 year after initial SRS (surgery, SRS, laser interstitial thermal therapy, or whole brain radio-therapy).

SECONDARY OUTCOMES:
Intracranial objective response rate | 2 years
  Determine the intracranial objective response rate, as measured by Response Assessment in Neuro-Oncology (RANO) criteria
Systemic objective response rate | 2 years
  Determine the systemic objective response rate, as measured by iRECIST criteria
Radiation necrosis-free survival at 1 year | 1 year
Overall survival | 2 years
  Determine the overall survival of patients with melanoma brain metastases treated with CA-4948 and pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Bently Doonan, MD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States